CLINICAL TRIAL: NCT01010490
Title: A Randomised Trial of Torsional Ultrasound Versus Longitudinal Ultrasound During Phacoemulsification of Age-related Cataracts: Comparison of Intra-operative Performance and Impact on Post-operative Endothelium Integrity
Brief Title: Outcomes of Phacoemulsification With Torsional Ultrasound
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Shetal Raj, Raghudeep eye clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-009
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Cataract
Keywords: PACHYMETRY; CELL LOSS; SAFETY; EFFICACY; PHACOEMULSIFICATION; Intraoperative complications; CLOCK TIME; FLUID USED; CORNEAL THICKNESS; ENDOTHELIUM CELL LOSS
MeSH Terms: conditions — Cataract; Intraoperative Complications | interventions — methylacetylene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Torsional ultrasound (Experimental): Torsional ultrasound with the INFINITI phacoemulsification system (Alcon Lab, USA)
  Interventions: Procedure: Torsional ultrasound (INFINITI, Alcon, USA)
- Longitudinal ultrasound (INFINITI) (Active Comparator): Longitudinal ultrasound with the INFINITI phacomachine (Alcon Lab, USA)
  Interventions: Procedure: Longitudinal U/S (Infiniti system, Alcon, USA)
- Longitudinal ultrasound (LEGACY) (Active Comparator): Longitudinal ultrasound with the LEGACY phacomachine (Alcon Lab, USA)
  Interventions: Procedure: Longitudinal U/S (LEGACY 20000, Alcon, USA)

INTERVENTIONS:
Procedure: Torsional ultrasound (INFINITI, Alcon, USA) — Comparison of inta-operative efficacy and safety
  Other Names: OZIL technology
  Arms: Torsional ultrasound
Procedure: Longitudinal U/S (Infiniti system, Alcon, USA) — comparison of efficacy and safety
  Other Names: traditional ultrasound
  Arms: Longitudinal ultrasound (INFINITI)
Procedure: Longitudinal U/S (LEGACY 20000, Alcon, USA) — Interrupted energy modality
  Other Names: Traditional U/S
  Arms: Longitudinal ultrasound (LEGACY)

SUMMARY:
To determine the differences in intra-operative complications, surgical duration, fluid usage, corneal thickness and endothelium cell density in eyes undergoing microcoaxial phacoemulsification (MCP) either with Torsional or longitudinal ultrasound during the surgery and at post-operative day 1, 1 month and 3 months.

DETAILED DESCRIPTION:
Introduced in mid 2006, torsional ultrasound (OZil, Infiniti Vision System, Alcon Laboratories, Texas, USA) uses rotational oscillations at ultrasonic frequencies to emulsify cataractous lens material in a seamless cutting motion from a tip that oscillates laterally. The side-to-side movement of the phaco tip produces minimal repulsion of lens material from the phaco tip resulting in improved followability. Clinically this translates into more effective lens removal with torsional phaco in comparison to the conventional ultrasound mode.to test this in a clinical scenario we undertook this study.

ELIGIBILITY:
Inclusion Criteria:

* patients 55 years and older with a senile cataract grades 1 to 5 nuclear sclerosis based on Emery's classification,
* endothelial cell density > 1500 cells/mm2,
* anterior chamber depth > 2.4 mm, and
* a dilated pupil > 7 mm.

Exclusion Criteria:

* eyes with pseudoexfoliation,
* mature, traumatic, or complicated cataracts,
* history of previous intra-ocular surgery, glaucoma, uveitis, and
* patients who were unable to comply with follow-up examinations.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Intra-operative complications, surgical clock time in minutes (SCT), fluid volume in ml(FV), and central corneal thickness in µm (CCT) on day 1 and months 1 and 3, and endothelial cell density (ECD) at 3 months. | 3 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: shetal m raj, ms, Principal Investigator — Iladevi Cataract and IOL Research Center
Locations (1):
- Raghudeep eye clinic, Ahmedabad, Gujarat, India

REFERENCES:
- [Result] Liu Y, Zeng M, Liu X, Luo L, Yuan Z, Xia Y, Zeng Y. Torsional mode versus conventional ultrasound mode phacoemulsification: randomized comparative clinical study. J Cataract Refract Surg. 2007 Feb;33(2):287-92. doi: 10.1016/j.jcrs.2006.10.044. PMID 17276271